CLINICAL TRIAL: NCT03668639
Title: A Study to Investigate the Safety and Antiemetic Efficacy of Akynzeo Plus Dexamethasone in Patients Receiving Concomitant Chemo-radiotherapy With Weekly Cisplatin for at Least Five Weeks
Brief Title: Safety and Antiemetic Efficacy of Akynzeo Plus Dexamethasone During Radiotherapy and Concomitant Weekly Cisplatin
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christina Ruhlmann (Other)
Collaborators: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor-Investigator, Christina Ruhlmann, Principal investigator, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DANGER-emesis
Record Dates: First submitted 2018-01-28; First posted 2018-09-12 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Chemotherapy-induced Nausea and Vomiting; Adverse Event; Cervical Cancer
MeSH Terms: conditions — Vomiting; Uterine Cervical Neoplasms | interventions — netupitant, palosentron drug combination; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Akynzeo plus dexamethasone (Other): Akynzeo (capsule 300mg/0.5mg) Day 1 plus dexamethasone 12 mg Day 1, 8 mg Day 2-3, and 4 mg Day 4 to be administered weekly for five weeks.
  Interventions: Drug: Akynzeo; Drug: Dexamethasone

INTERVENTIONS:
Drug: Akynzeo — Weekly administration of akynzeo for five weeks.
Drug: Dexamethasone — Weekly administration of dexamethasone 12 mg Day 1, 8 mg Day 2-3, and 4 mg Day 4 for five weeks.

SUMMARY:
This is a multicentre, single-arm, phase II study to investigate the safety and antiemetic efficacy of Akynzeo (a fixed dose combination of palonosetron and netupitant) plus dexamethasone in patients receiving concomitant chemo-radiotherapy with weekly cisplatin for at least five weeks.

DETAILED DESCRIPTION:
Akynzeo contains a combination of the neurokinin-1 receptor antagonist netupitant and the serotonin receptor antagonist palonosetron. Akynzeo is approved as antiemetic prophylaxis in patients receiving high emetogenic chemotherapy e.g. high dose cisplatin administered every three weeks.

From a previous clinical trial (GAND-emesis trial) we know that patients receiving radiotherapy and concomitant weekly cisplatin 40 mg/m2 are better protected against nausea and vomiting when a triplet antiemetic prophylaxis (neurokinin-1 receptor antagonist, serotonin receptor antagonist, and corticosteroid) is applied.

In the Akynzeo phase III clinical trials, Akynzeo was administered every three weeks. The neurokinin-1 receptor antagonist, netupitant, has a long plasma half-life (approx. 90 hours), and theoretically the drug could accumulate when administered on a weekly basis.

The DANGER-emesis trial is designed to collect safety and efficacy data in patients receiving Akynzeo weekly as antiemetic prophylaxis in combination with dexamethasone in patients treated for cervical cancer with radiotherapy and concomitant weekly cisplatin 40 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of cervical cancer.
2. The patient understands the nature and purpose of this study and the study procedures and has signed informed consent.
3. The patient is aged ≥ 18 years.
4. The patient must be both chemo- and radiotherapy (RT) naïve. NB: previously low voltage RT or electron RT for non-melanoma skin cancers is allowed.
5. The patient is scheduled to receive fractionated radiotherapy and concomitant weekly cisplatin at a dose of ≥ 40 mg/m2 for at least five weeks.
6. Brachy therapy is scheduled to be initiated after the third cycle of weekly cisplatin, and preferentially after the fifth week of treatment.
7. Chemotherapy with an emetic risk potential of minimal or mild (up to 30%) is allowed on days 1-4 (see ref. 14).
8. The patient has a WHO Performance Status of ≤ 2.
9. Hematologic and metabolic status must be adequate for receiving weekly cisplatin in a dose of ≥ 40 mg/m2, and meet the following criteria:

   * Total neutrophils ≥ 1500/mm3 (Standard units : ≥1.5 x 109/L)
   * Platelets ≥ 100,000/mm3 (Standard units: ≥100.0 x 109/L)
   * Bilirubin ≤ 1.5 x ULN (Upper Limits of Normal)
   * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 x ULN
   * GFR ≥ 50 ml/min
10. The patient is able to read, understand, and complete questionnaires and daily components of the Patient Diary for each study cycle.
11. For patients of childbearing potential, urine human chorionic gonadotropin (hCG) (urine dipstick pregnancy test) or blood hCG results must be negative at screening, and these patients must agree to one of the following methods of contraception:

    * Hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release).
    * Male partner who is sterile prior to the patient's entry into the study and is the sole sexual partner for that patient.
    * Complete abstinence from intercourse for two weeks before study entry and throughout the study period plus a period after the trial to account for elimination of the drug (minimum of eight days). Abstinence is only an acceptable contraception form, when it reflects the usual and preferred lifestyle of the patient.

Exclusion Criteria:

1. The patient has a current malignant diagnosis other than cervical cancer, with exception of non-melanoma skin cancers.
2. The patient is pregnant or lactating.
3. The patient has experienced emesis (i.e., vomiting and/or retching) or clinically significant nausea (defined as nausea graded as moderate or severe) in the 24 hours preceding the first dose of study medication.
4. The patient has a history active peptic ulcer disease, gastrointestinal obstruction, gastrointestinal carcinoma, increased intracranial pressure, hypercalcemia, or any uncontrolled medical condition (other than malignancy) which in the opinion of the Investigator may confound the results of the study, represent another potential etiology for emesis and nausea (other than CINV/RINV) or pose an unwarranted risk to the patient.
5. The patient has a known hypersensitivity or contraindication to palonosetron, another 5-HT3 receptor antagonist, dexamethasone, or netupitant.
6. The patient has previously received an NK1 receptor antagonist.
7. The patient has received an investigational drug in the previous 30 days or is scheduled to receive any investigational drug during the study period.
8. The patient has taken/received any medication of moderate or high emetogenic potential within the 48 hours prior to the first dose of study medications. Opiate drugs for cancer pain will be permitted if the patient has been on a stable dose and has not experienced emesis or clinically significant nausea from the narcotics in the 24 hours preceding the first dose of study medication.
9. The patient has taken/received any medication with known or potential antiemetic activity within the 24-hour period prior to receiving study drugs. This includes, but is not limited to:

   * 5-HT3 receptor antagonists (e.g., ondansetron, granisetron, dolasetron, tropisetron, ramosetron). Palonosetron is not permitted within 7 days prior to receiving study drugs.
   * Benzamide / benzamide derivatives (e.g., metoclopramide, alizapride).
   * Benzodiazepines (except if the patient is receiving such medication for sleep or anxiety and has been on a stable dose for at least seven days prior to the first dose of study medications).
   * Phenothiazines (e.g., prochlorperazine, promethazine, metopimazine, fluphenazine, perphenazine, thiethylperazine, chlorpromazine).
   * Butyrophenone (e.g., haloperidol, droperidol).
   * Corticosteroids (e.g., dexamethasone, methylprednisolone, prednisolone; with the exception of topical steroids for skin disorders, inhaled steroids for respiratory disorders).
   * Anticholinergics (e.g., scopolamine).
   * Antihistamines (e.g., cyclizine, hydroxyzine, diphenhydramine).
   * Domperidone.
   * Cannabinoids.
   * Mirtazapine.
   * Olanzapine.
10. The patient has taken/received strong or moderate inhibitors of CYP3A4 within seven (7) days prior to administration of study drugs (see Section 10.3.1., "Inhibitors of CYP3A4").
11. The patient has taken/received inducers of CYP3A4 within thirty (30) days prior to the administration of study drugs (see Section 10.3.2., "Inducers of CYP3A4").

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with cervical cancer.
Enrollment: 80 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Safety of weekly administration of Akynzeo measured by incidence of treatment-emergent adverse events | Five weeks.
  Measurement of incidence of treatment-emergent adverse events.
Efficacy of weekly administration of Akynzeo measured by incidence of nausea and vomiting and use of rescue antiemetics | Five weeks.
  Measurement of incidence of nausea and vomiting and use of rescue antiemetics.

SECONDARY OUTCOMES:
Complete response in terms of the proportion of subjects with complete response | Five days and five weeks.
  To investigate Akynzeo and dexamethasone in terms of the proportion of subjects with complete response (defined as no vomits, no dry retches and no need for rescue medication) in the 5 days and the 35 days following initiation of fractionated radiotherapy and concomitant weekly cisplatin at a dose of ≥ 40 mg/m2.
No significant nausea in terms of the proportion of subjects with no significant nausea | Five days and five weeks.
  To investigate Akynzeo and dexamethasone in terms of the proportion of subjects with no significant nausea (none or mild nausea) in the 5 days and the 35 days following initiation of fractionated radiotherapy and concomitant weekly cisplatin at a dose of ≥ 40 mg/m2.
No nausea in terms of the proportion of subjects with no nausea | Five days and five weeks.
  To investigate Akynzeo and dexamethasone in terms of the proportion of subjects with no nausea in the 5 days and the 35 days following initiation of fractionated radiotherapy and concomitant weekly cisplatin at a dose of ≥ 40 mg/m2.
Time to first emetic episode | Five weeks.
  To investigate Akynzeo and dexamethasone in terms of time to first emetic episode.

CONTACTS AND LOCATIONS:
Overall Officials: Christina H. Ruhlmann, MD, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Oncology, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Detlefsen SS, Andersen DS, Knudsen AO, Nottrup TJ, Moller S, Nyvang GB, Jorgensen TL, Herrstedt J, Ruhlmann CH. Safety and antiemetic efficacy of weekly administration of netupitant/palonosetron plus dexamethasone during 5 weeks of concomitant chemo-radiotherapy-the DANGER-emesis study. Support Care Cancer. 2025 May 28;33(6):509. doi: 10.1007/s00520-025-09573-9. PMID 40437122